CLINICAL TRIAL: NCT00070915
Title: Relaxation-Related CAM Therapies for Chronic Back Pain
Brief Title: Massage, Meditation, and Tai Chi for Chronic Lower Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: R01AT000606-01 (NIH); R01AT000606-01 (NIH)
Record Dates: First submitted 2003-10-09; First posted 2003-10-13 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Tai Ji; Massage

INTERVENTIONS:
Behavioral: Tai chi
Behavioral: Mindfulness-based Stress Reduction program
Procedure: Therapeutic massage

SUMMARY:
This clinical trial is a preliminary study designed to prepare for a full-scale, randomized clinical trial of the effectiveness of tai chi, mediation, and therapeutic massage for chronic lower back pain in adults.

DETAILED DESCRIPTION:
Despite the common use of complementary and alternative therapies for back pain, little is known about how such therapies compare with each other or with conventional medical therapies in terms of effectiveness and cost. This study will lay the groundwork for a full-scale trial that will evaluate the relative effectiveness and costs of three promising relaxation-related techniques (massage, tai chi, and meditation) that are appropriate for both younger and older adults with chronic lower back pain. The pilot study will identify and resolve unanticipated problems and estimate the sample sizes required for an adequately-powered, full-scale trial.

Participants with chronic lower back pain will be randomly assigned to one of the following groups: tai chi, massage, meditation, or continued usual care (control group). The participants assigned to each intervention will be divided equally between persons under and over age 65.

ELIGIBILITY:
Inclusion Criteria

* Chronic lower back pain

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120
Dates: Start 2000-09; Study Completion 2003-06

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C. Cherkin, Principal Investigator — Center for Health Studies